CLINICAL TRIAL: NCT02281994
Title: Safety and Efficacy of Pulsed Electromagnetic Fields (Cervical-Stim®) as an Adjunct to Enhance Union in Conservatively Treated Type II Fractures of the Odontoid Process
Brief Title: Odontoid Fracture Study Treated With Pulsed Electromagnetic Fields
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-1402ODFX
Record Dates: First submitted 2014-10-26; First posted 2014-11-04 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Odontoid Fracture Type II
Keywords: PEMF; odontoid fracture; IDE; prospective

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active PEMF (Active Comparator): Active device emits Pulsed Electromagnetic Field (PEMF)
  Interventions: Device: Pulsed Electromagnetic Feld (PEMF) Orthofix Cervical-Stim Model 2205OD
- Control/no PEMF (Placebo Comparator): control/placebo device does not emit Pulsed Electromagnetic Field (PEMF)
  Interventions: Device: Pulsed Electromagnetic Feld (PEMF) Orthofix Cervical-Stim Model 2205OD

INTERVENTIONS:
Device: Pulsed Electromagnetic Feld (PEMF) Orthofix Cervical-Stim Model 2205OD — Active devices emit PEMF signal; control devices do not emit PEMF signal.

SUMMARY:
The hypothesis of this study is that PEMF treatment will improve odontoid fracture healing, compared with standard conservative care, in subjects 50 years of age and over diagnosed with Type II odontoid fractures, and this effect will be evident by 6 months post-injury. Subjects will be assessed for the presence of a Type II odontoid fracture by X-ray, MRI and CT scan. Subjects meeting eligibility criteria will be randomized in a 2:1 ratio (active: placebo control) to either the active or control device for 4 hours a day for 6 months. X-rays will be collected at 6 weeks, and at 3, 6 and 12 months to assess the fracture healing process, with flexion-extension x-rays collected at 3, 6 and 12 months. A CT scan will be performed at 6 months to confirm healing. Quality of Life measures (SF-36, VAS neck pain scale, NDI) will be collected at all visits (6 weeks, 3, 6 and 12 months). Study subjects will receive either an active Orthofix Cervical-Stim Model 2205OD or an inactive (placebo) Orthofix Cervical-Stim Model 2205OD device.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 50 years of age or older at the time of consent
* Subject must have radiographic evidence (x-ray , MRI and CT scan) of a Type II odontoid fracture
* Subject must have MRI evidence that the fracture occurred within 30 days of study enrollment
* Subject must have VAS neck pain score of greater than 4 (>4)
* Subject must have radiographic evidence that the fracture is displaced ≤ 5 mm in any direction and/or have a fracture gap of ≤ 3 mm due to angulation
* Subject must use a rigid cervical collar (Miami J, Philadelphia or Aspen) for a minimum of three months post-injury
* Subject must have a DEXA scan within 6 months prior to enrollment (can be done within one week of baseline visit)
* Subject must be willing and able to follow all study procedures and return for all study visits
* Subject must be willing to sign an Informed Consent Document

Exclusion Criteria:

* Subject has undergone systematic administration, within 30 days prior to the fracture, of any type of corticosteroid, antineoplastic, immunostimulation or immunosuppressive agents
* Subject is on chronic anticoagulation, or has a bleeding disorder
* Subject is pregnant, nursing or plans to become pregnant during the study
* Subject has a chronic Type II odontoid fracture that occurred more than 21 days prior to enrollment
* Subject has a Type II odontoid fracture displaced >5 mm
* Subject has a mental or physical condition that would prevent him from complying with the study protocol, including the physician obtaining an accurate neurologic exam
* Subject was recommended for surgery to treat the fracture but subject refused surgery
* Subject is a prisoner
* Subject has participated in another clinical trial within the last 90 days

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change over time of VAS pain | Baseline, 6 week, 3 month, 6 month, 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Paul Arnold, MD, Principal Investigator — The University of Kansas Hospital; Wellington Hsu, MD, Principal Investigator — Northwestern University; Zachary Ray, MD, Principal Investigator — Washington University School of Medicine; Khalid Abbed, MD, Principal Investigator — Yale University; Joshua Ammerman, MD, Principal Investigator — Washington Neurosurgical Associates; Jung Yoo, MD, Principal Investigator — Oregon Health and Science University; Kelly Banagan, MD, Principal Investigator — University of Maryland, College Park; Kee Kim, MD, Principal Investigator — UC Davis; Sanjay Dhall, MD, Principal Investigator — UC San Francisco; Amir Vokshoor, MD, Principal Investigator — DISC Sports and Spine Center